CLINICAL TRIAL: NCT05679570
Title: Satralizumab,an Anti-IL-6 Receptor Antibody, in the Treatment of Pulmonary Arterial Hypertension; Safety and Efficacy Evaluation in Japan -Multicenter, Investigator-sponsored Trial-
Brief Title: Satralizumab in the Treatment of Pulmonary Arterial Hypertension (SATISFY-JP Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International University of Health and Welfare (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Keio University (Other); Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-001-SA237; jRCT2031210626 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2022-12-04; First posted 2023-01-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — satralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Satralizumab （Genetical Recombination） (Experimental)
  Interventions: Drug: Satralizumab (Genetical Recombination)

INTERVENTIONS:
Drug: Satralizumab (Genetical Recombination) — Efficacy Evaluation Period:
  The study drug will be administered at a dose of 120 mg subcutaneously at initial, 2-week, 4-week, and 4-week intervals thereafter. Efficacy will be assessed after 24 weeks of study drug administration. Subjects who demonstrate efficacy and wish to continue treatment will receive the study drug for 24 weeks and moving to the continuous treatment period. In all other cases, the study will be terminated after 24 weeks of the efficacy evaluation period without the administration of study drug.
  Continuation Dosing Period[1]:
  Subjects who demonstrate efficacy during the efficacy evaluation period and wish to continue will receive continued 28 weeks (52 weeks total) treatment with satralizumab.
  Continuation Dosing Period[2]:
  Subjects completed continuation dosing period[1], clinically capable of continued administration, and wish to continue will receive continued treatment with satralizumab until the end of this study period.

SUMMARY:
Examine the efficacy of satralizumab in patients with pulmonary arterial hypertension (PAH) with immune-responsive phenotype serum interleukin-6 (IL-6) ≥ 2.73 pg/mL who have an inadequate response to existing drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age at the time of consent acquisition is between 20 and 80 years old.
2. Patients who have been diagnosed with pulmonary arterial hypertension (PAH) and fall into one of the following among the first group of the clinical classification of pulmonary hypertension (Nice Classification, 2018) Idiopathic pulmonary arterial hypertension (IPAH) Hereditary pulmonary arterial hypertension (HPAH) Drug/toxin-induced pulmonary arterial hypertension Pulmonary arterial hypertension associated with connective tissue disease Pulmonary arterial hypertension associated with congenital heart disease (only after repair surgery)
3. Patients in the World Health Organization (WHO) Functional Classification (FC) I, II, or III.
4. Patients with immune responsive-phenotype
5. Patients with a 6-minute walking distance of 150 to 600 meters at screening.
6. Patients whose resting hemodynamic values within 30 days prior to enrollment meet all of the following Mean pulmonary artery pressure (mPAP) is 25 mmHg or higher PVR is higher than 4 Wood units
7. Patients who are using up to three PAH drugs and have not changed the dosage and administration for at least 90 days prior to enrollment
8. Patients who are receiving home oxygen therapy under the same conditions for at least 30 days prior to enrollment
9. Patients who have given written consent for the study

Exclusion Criteria:

1. Patients with a history of severe allergy to any of the components of the study drug.
2. Patients who have received IL-6 inhibitors (tocilizumab, sarilumab, etc.) in the past or are currently receiving them at the time of screening.
3. Patients with infectious diseases such as pneumonia or tuberculosis during the screening period.
4. Patients with pulmonary artery wedge pressure (PAWP) greater than 15 mmHg on the last right heart catheterization performed during the screening period.
5. Patients who are using epoprostenol (intravenous) or treprostinil (intravenous or subcutaneous) and cannot discontinue.
6. Patients who are currently participating in other clinical trials or clinical studies. Or, patients who have participated in other clinical trials/trials prior to participation in this study and whose adverse events, if any, have occurred during the period of participation and have not been confirmed to have resolved or stabilized
7. Pregnant women or lactating patients.
8. Patients who are unable to consent to contraception from the time of obtaining consent until at least 3 months after the last dose of the study drug
9. Patients who have received a live vaccine within 6 weeks prior to enrollment
10. Patients who are positive for HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, HBs antigen, or HCV antibody.
11. Patients with active or recurrent bacterial, viral, fungal, or mycobacterial infections, or with other infectious diseases
12. Patients who have been hospitalized or developed an infection requiring intravenous administration of an infectious agent within 4 weeks prior to the baseline visit or an infection requiring oral administration of an infectious agent within 2 weeks prior to the baseline visit.
13. Patients who are receiving steroids at a dose higher than 10 mg/day of prednisone (PSL) equivalent.
14. Patients with a history of malignancy, including solid tumors, hematologic malignancies, and intraepithelial carcinomas, within the past 5 years.
15. Patients who are judged to lack the capacity to consent.
16. Other patients who are judged by the investigator to be unsuitable for the study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in total pulmonary vascular resistance (PVR) from baseline to 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
The change in the 6-minute walking distance from baseline to 24 weeks. | 24 weeks
Comparison of the percent change in PVR from baseline to 24 weeks between the satralizumab group in this study and an external control group (selected from patients enrolled in JAPHR). | 24 weeks
Number of participants with treatment-related adverse events as assessed by MedDRA and changes in general laboratory test values. | 52 weeks, beyond 52 weeks(1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Yuichi Tamura, Study Chair — International University of Health and Welfare
Locations (9):
- Japan (9):
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Kobe University Hospital, Kobe
  - Kurume University Hospital, Kurume
  - Kyorin University Hospital, Mitaka
  - Nagoya University Hospital, Nagoya
  - Hokkaido University Hospital, Sapporo
  - International University of Health and Welfare Mita Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No